CLINICAL TRIAL: NCT01684592
Title: Phone-Based Postpartum Continuing Care: Smoking Cessation Beginning in Pregnancy
Brief Title: Phone-Based Postpartum Continuing Care for Smoking Cessation
Acronym: PPCC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Battelle Memorial Institute (Other)
Collaborators: University of Maryland (Other); Chestnut Health Systems (Other)
Responsible Party: Principal Investigator, Victoria H. Coleman-Cowger, Principal Research Scientist, Battelle Memorial Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1R34DA032683-01A1 (NIH)
Record Dates: First submitted 2012-09-11; First posted 2012-09-13 (Estimated); Results first posted 2018-03-13 (Actual); Last update posted 2018-03-13 (Actual); Status verified 2018-02

CONDITIONS: Smoking Cessation; Pregnancy
Keywords: smoking cessation; relapse prevention; pregnancy; postpartum
MeSH Terms: conditions — Smoking Cessation | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard care (Active Comparator): Standard care for smokers during pregnancy and referral to 24/7 quitline postpartum (passive)
  Interventions: Behavioral: Standard care
- Standard care plus PPCC (Experimental): Standard care for smoking during pregnancy and proactive phone-based postpartum continuing care (PPCC) for 6 months postpartum
  Interventions: Behavioral: Phone-based postpartum continuing care; Behavioral: Standard care

INTERVENTIONS:
Behavioral: Phone-based postpartum continuing care — PPCC Counselors will make initial contact with participants in the experimental group at 36 weeks gestation (i.e., one week prior to full-term), will call again within one week after the baby's birth, and eight additional times over the course of the first six months postpartum. The PPCC protocol will be developed based on the 5 A's (standard of care during pregnancy) and the Recovery Management Checkup model where relapse is expected and efforts are made to take a more proactive approach to identify women who are having cravings or have relapsed and re-intervene with them as soon as possible to assist them in regaining smoking abstinence. Women in the experimental group will also have the option of calling the PPCC line 24 hours a day, 7 days a week.
  Other Names: PPCC
  Arms: Standard care plus PPCC
Behavioral: Standard care — All women will receive the standard of care approach (5 A's and referral to a 24/7 quit line postpartum) from MWC during pregnancy. The 5 A's brief intervention was modified by American College of Obstetricians and Gynecologists (ACOG) for use with pregnant women and is recommended to help pregnant women quit smoking. It includes the following steps: Ask about tobacco use, Advise to quit, Assess willingness to make a quit attempt, Assist in quit attempt, and Arrange follow-up.

SUMMARY:
Smoking is a leading cause of death and other negative health outcomes. While a high percentage of women quit smoking during pregnancy, the majority relapse in the first 6 months postpartum. We propose developing and pilot testing a phone-based postpartum continuing care (PPCC) protocol based on existing evidence-based approaches to increase smoking cessation, reduce relapse, increase early re-intervention, and reduce infant exposure to environmental tobacco smoke in the postpartum period.

DETAILED DESCRIPTION:
The large majority of women who quit smoking during pregnancy relapse in the first six months postpartum, highlighting a need for effective postpartum continuing care that supports women through the challenging postpartum period when stress is high and motivation to stay quit may decline. Existing relapse prevention interventions (typically delivered during pregnancy) have been found to be of little benefit during the postpartum period, suggesting the need for a more formal continuing care approach. Phone-based protocols for smoking cessation have been widely disseminated and effective because they address the need for flexible access, but are passive and not typically utilized by women in the postpartum period.

The proposed pilot study will develop and test a Phone-based Postpartum Continuing Care (PPCC) model that draws from existing evidence-based protocols--the 5 A's and Recovery Management Checkups (RMC)-- shown to be effective with other populations. The experimental PPCC will reinforce the importance of abstinence, relapse prevention, and reduced smoking through proactive re-intervention (i.e., RMC) with the 5 A's at times when postpartum women are more likely to relapse, and provide education and monitoring of the infant's direct and indirect exposure to nicotine through breastfeeding and secondhand smoke. We will evaluate PPCC's effectiveness relative to a passive referral to a 24/7 hotline, which is current standard care.

Approximately one hundred thirty women in their first or second trimester of pregnancy who were nicotine-dependent in the past year, currently smoke, or quit within the past 90 days will be recruited at their first prenatal appointment at the Maryland Women's Center (MWC) in Baltimore, Maryland. All women will receive the clinic's standard of care for smoking cessation--the 5 A's --during pregnancy from their physician. Half will be randomly assigned to an experimental group getting PPCC for 6 months postpartum and half to a control group receiving only a referral to a passive 24/7 state quit line postpartum. It is expected that in the 6 months following childbirth women in the experimental PPCC (relative to those in the control group) will: a) smoke fewer cigarettes, b) smoke fewer days, c) go longer before postpartum relapse, d) have less time between relapse and talking to a health professional about smoking, e) have less time between relapse and resumption of abstinence , f) smoke fewer times while breastfeeding, g) smoke fewer times while in the same room as the infant, and h) reduce their infant's cotinine levels.

The aims of this pilot project are to develop PPCC from existing evidence-based approaches, demonstrate the feasibility of implementing the PPCC intervention with at least 80% compliance and at least 80% follow-up at each wave, and evaluate the effect size associated with receiving standard care vs. standard care + PPCC in order to understand the promise of and appropriate power required for a larger clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* first or second trimester of pregnancy
* age 18 or older
* self-reported tobacco use in the past 90 days or nicotine-dependence in the past year

Exclusion Criteria:

* intend to terminate their pregnancy
* intend to move out of the city within the next 12 months
* are unable to provide informed consent and participate in English

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2012-10; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Victoria H Coleman-Cowger, PhD, Principal Investigator — Battelle Memorial Institute; Katrina Mark, MD, Study Director — University of Maryland, Baltimore
Locations (2):
- United States (2):
  - Chestnut Global Partners, Bloomington, Illinois
  - Maryland Women's Center, Baltimore, Maryland

IPD SHARING:
Plan to Share IPD: No
Researchers may request de-identified aggregate data in 2017 via email from the PI of record by submitting a formal request with desired variables.

REFERENCES:
- [Background] Coleman-Cowger VH. Smoking cessation intervention for pregnant women: a call for extension to the postpartum period. Matern Child Health J. 2012 Jul;16(5):937-40. doi: 10.1007/s10995-011-0837-2. PMID 21710186

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The sample was drawn from a population of low-income pregnant women attending their first prenatal visit at an obstetrics clinic in Baltimore, MD. In total, 790 women (i.e., smokers and non-smokers) were assessed for eligibility from March-December 2013, with 180 meeting eligibility criteria. Of those screened, 130 participants were enrolled.
Pre-assignment Details: Randomization occurred at week 26 gestation, after intake data was collected.
Groups:
- Standard Care: Standard care for smokers during pregnancy and referral to 24/7 quitline postpartum (passive)
  Standard care: All women will receive the standard of care approach (5 A's and referral to a 24/7 quit line postpartum) from Maryland Women's Clinic (MWC) during pregnancy. The 5 A's brief intervention was modified by the American College of Obstetricians and Gynecologists (ACOG) for use with pregnant women and is recommended to help pregnant women quit smoking. It includes the following steps: Ask about tobacco use, Advise to quit, Assess willingness to make a quit attempt, Assist in quit attempt, and Arrange follow-up.
Period: Overall Study
Arm/Group | Standard Care | Standard Care Plus PPCC
Started (No intake data for two participants, thus only 128 were randomized.) | 64 | 64
Completed | 38 | 40
Not Completed | 26 | 24

BASELINE CHARACTERISTICS:
Groups:
- Standard Care: Standard care for smokers during pregnancy and referral to 24/7 quitline postpartum (passive)
  Standard care: All women will receive the standard of care approach (5 A's and referral to a 24/7 quit line postpartum) from MWC during pregnancy. The 5 A's brief intervention was modified by ACOG for use with pregnant women and is recommended to help pregnant women quit smoking. It includes the following steps: Ask about tobacco use, Advise to quit, Assess willingness to make a quit attempt, Assist in quit attempt, and Arrange follow-up.
- Total: Total of all reporting groups
Arm/Group | Standard Care | Standard Care Plus PPCC | Total
Number analyzed (Participants) | 64 | 64 | 128
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.6 (4.7) | 26.3 (5.3) | 26.0 (5.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 64 | 64 | 128
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 53 | 50 | 103
  White | 7 | 13 | 20
  More than one race | 4 | 1 | 5
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 64 | 64 | 128

OUTCOME MEASURES:

1. Primary Outcome: Number of Tobacco Products Per Day
Description: Self-reported number of tobacco products smoked per day
Time Frame: 6 months postpartum
Measure: Mean (95% Confidence Interval); unit: tobacco products
Arm/Group | Standard Care | Standard Care Plus PPCC
Number analyzed (Participants) | 64 | 64
tobacco products | 6.4 [4 to 8] | 6.9 [5 to 9]

2. Secondary Outcome: Number of Tobacco Products Per Day
Description: Self-reported number of tobacco products smoked per day
Time Frame: 3 months postpartum
Measure: Mean (95% Confidence Interval); unit: tobacco products
Arm/Group | Standard Care | Standard Care Plus PPCC
Number analyzed (Participants) | 64 | 64
tobacco products | 7.1 [5 to 9] | 7.9 [6 to 10]

3. Secondary Outcome: Past 90-day Tobacco Use
Description: Self-reported number of days smoked in past 90 days
Time Frame: 3 months postpartum
Measure: Mean (95% Confidence Interval); unit: days
Arm/Group | Standard Care | Standard Care Plus PPCC
Number analyzed (Participants) | 64 | 64
days | 60.7 [49 to 72] | 57.5 [45 to 70]

4. Secondary Outcome: Past 90-day Tobacco Use
Description: Self-reported number of days smoked tobacco in past 90 days.
Time Frame: 6 months postpartum
Measure: Mean (95% Confidence Interval); unit: days
Arm/Group | Standard Care | Standard Care Plus PPCC
Number analyzed (Participants) | 64 | 64
days | 59.2 [47 to 71] | 55.3 [41 to 69]

5. Secondary Outcome: Times Mother Smoked While Breastfeeding
Description: Based on the days of smoking while breastfeeding (or within 30 minutes of breastfeeding) times the frequency of use on day.
Time Frame: Baby's birth to 6 months postpartum
Population: Only 7 women reported having breastfed at 6 month postpartum
Measure: Mean (Standard Deviation); unit: times smoked in past 90 days
Arm/Group | Standard Care | Standard Care Plus PPCC
Number analyzed (Participants) | 3 | 4
times smoked in past 90 days | 7.13 (4.6) | 0 (0)

6. Secondary Outcome: Times Mother Smoked in the Room With Infant
Description: Based on the number of days of smoking in the same room with infant in the past 90.
Time Frame: Baby's birth to 6 months postpartum
Population: Only current smokers responded to this question
Measure: Mean (Standard Deviation); unit: number of days smoked
Arm/Group | Standard Care | Standard Care Plus PPCC
Number analyzed (Participants) | 33 | 36
number of days smoked | .70 (3.5) | .06 (.3)

7. Secondary Outcome: NicCheck Test Results for Cotinine Level From Infant Urine
Description: Infant urine was collected at 6 months postpartum using the "cotton roll" method of urine collection. Cotinine was measured with NicCheck I Test Strips that determine the urinary concentration of nicotine and its metabolites based on a colorimetric reaction. The test strip is dipped into participant's urine and changes color (varying shades of pink) in the presence of cotinine. Cotinine level is determined by matching the test strip with a color chart provided by the manufacturer. The intensity of color on the strip at the end of 15 minutes may be compared to those on the color chart, to differentiate between "low" (score 1-6) versus "high" (score 7-14) nicotine consumption. Absence of a color is considered a negative result (score 0). Based on comparison with gas chromatography urine cotinine values, individuals with cotinine values of 200 ng/mL and above are classified as smokers.
Time Frame: 6 months postpartum
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Standard Care | Standard Care Plus PPCC
Number analyzed (Participants) | 38 | 40
units on a scale | 0 (0) | 0 (0)

ADVERSE EVENTS:
Arm/Group | Standard Care | Standard Care Plus PPCC
Serious Adverse Events (participants affected / at risk) | 5/64 | 0/64
Other Adverse Events (participants affected / at risk) | 0/64 | 0/64
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Care (N=64) | Standard Care Plus PPCC (N=64)
Miscarriage (Pregnancy, puerperium and perinatal conditions) | 5 (5) | 0 (0) — Five participants miscarried prior to randomization at week 26 but following study enrollment.

LIMITATIONS AND CAVEATS:
Trend of Experimental group being heavier smokers than Control group; Difficulty contacting participants for PPCC calls (limited delivery of intervention).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Informed Consent Form (2014-09-18): https://cdn.clinicaltrials.gov/large-docs/92/NCT01684592/ICF_000.pdf
  • Study Protocol (2013-05-28): https://cdn.clinicaltrials.gov/large-docs/92/NCT01684592/Prot_001.pdf